CLINICAL TRIAL: NCT05205525
Title: Aggressive Versus Restrictive Initiation of Antimicrobial Treatment in Critically Ill Patients With Suspected Ventilator Acquired Pneumonia Without Severity : a Before and After Observational Study
Brief Title: Delayed Antibiotic Therapy in Non-severe Ventilator Acquired Pneumonia (VAP)
Acronym: DELAVAP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR_DELAVAP
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Ventilator Associated Pneumonia; Critical Care; Antibiotic Therapy
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Restrictive antibiotic strategy
  Interventions: Other: Restrictive antibiotic strategy
- Aggressive (immediate) antibiotic strategy
  Interventions: Other: Aggressive antibiotic strategy

INTERVENTIONS:
Other: Restrictive antibiotic strategy — Implementation of a restrictive (delayed) antibiotic strategy in Ventilator Acquired Pneumonia suspicion without severity symptoms.
  Groups: Restrictive antibiotic strategy
Other: Aggressive antibiotic strategy — Implementation of an aggressive (immediate) antibiotic strategy in Ventilator Acquired Pneumonia suspicion without severity symptoms.
  Groups: Aggressive (immediate) antibiotic strategy

SUMMARY:
This retro-prospective monocentric observational study compare the impact of the implementation of a restrictive (delayed) versus aggressive (immediate) antibiotic strategy for Ventilator Acquired Pneumonia suspicion without severity symptoms.

DETAILED DESCRIPTION:
Ventilator acquired pneumonia (VAP) is the leading cause of nosocomial infection in intensive care patients, and has been associated with increased antibiotic consumption, increased morbidity and mortality. VAP diagnosis is difficult due to subjective or non-specific criteria. Delaying antibiotic treatment for VAP suspicion without severity symptoms raises question since the probability of VAP diagnosis, as well as the risk of delaying treatment, is very uncertain. It may nonetheless limit the environmental impact of antibiotic use which is a public health concern. We compared antibiotic sparing and patient outcome, before and after the implementation of a restrictive (delayed) antibiotic strategy versus an aggressive (immediate) antibiotic strategy in VAP suspicion without severity symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Under mechanical ventilation from more than 48 hours
* Suspected for a ventilator acquired pneumonia, requiring a distal pulmonary bacterial sample

Exclusion Criteria:

* New or worsening shock requiring vasopressor
* New or worsening severe hypoxemia (PaO2/FiO2<150 in FiO2≥60% and peep 10)
* Patient under veno-veinous extracorporeal membrane oxygenation
* Neutropenia <1G/L or immunosuppressive treatment (including corticosteroids >6 months or >0.5mg/kg/j)
* Disease (endocarditis, spondylodyscitis, deep abcedation…) requiring prolonged antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient under mechanical ventilation in intensive care with suspected ventilator acquired pneumonia
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
antibiotic-free days | 28 days
  antibiotic-free days until Day 28 of Intensive Care Units stay

SECONDARY OUTCOMES:
Mechanical ventilation free days | 28 days
  Mechanical ventilation free days during the first 28 days
Intensive care unit stay length | 28 days
Intensive care unit mortality | 28 days
Hospitality mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Nantes Hospital, Nantes, France